CLINICAL TRIAL: NCT00258674
Title: A Randomized Trial of Strategies to Improve Diabetes Care: Effectiveness and Costs of Physician Profiling and Care Coordination by a Diabetes Resource Nurse
Brief Title: Improving Diabetes Care:Effectiveness of Physician Profiling and Care Coordination by a Diabetes Resource Nurse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 000-113
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Care coordination; Case management; Physician profiling
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Medicare Claims Feedback (Active Comparator): Practices randomised to the Medicare Claims Feedback arm received period feedback on their performance on selected diabetes quality of care measures as reflected in the claims data for their diabetes patients.
  Interventions: Other: Medicare Claims Feedback
- Medicare Claims+Medical Record Feedback (Experimental): Practices randomised to the Medicare Claims + Medical Record Review Feedback arm received periodic feedback on their performance on selected diabetes quality of care measures as reflected in both the Medicare claims for the diabetes patients AND review/audit of their diabetes patients' medical records.
  Interventions: Other: Medicare Claims Feedback; Other: Medical Record Review
- Medicare Claims+Medical Chart Review+DRN (Experimental): In addition to the performance data from both Medicare Claims data and from review of patients' medical records, practices randomised to the Medicare Claims + Medical Record review + Diabetes Resource Nurse (DRN) had a diabetes resource nurse assigned to them, who was available to provide diabetes education and care-coordination type services for their diabetes patients.
  Interventions: Other: Medicare Claims Feedback; Other: Medical Record Review; Other: Diabetes Resource Nurse

INTERVENTIONS:
Other: Medicare Claims Feedback — Physician practices received periodic feedback on their performance on selected diabetes quality of care measures as reflected by the Medicare claims data for their patients.
Other: Medical Record Review — Physician practices received period feedback on their performance on selected diabetes quality of care measures, as reflected by data collected from their patients' medical records. These data were compiled by trained nurse abstractors using a standardized data collection tool developed for this study.
  Arms: Medicare Claims+Medical Chart Review+DRN; Medicare Claims+Medical Record Feedback
Other: Diabetes Resource Nurse — Diabetes Resource Nurses (DRNs) were registered nurses with 3-5 years of experience as certified diabetes educations who performed initial patient assessments, developed plans of care, administered screening tools, and monitored clinical outcomes. Physicians at the practices randomised to this intervention had could access the DRN's services for their diabetes patients, but neither physicians nor patients had to take advantage of this resource.
  Arms: Medicare Claims+Medical Chart Review+DRN

SUMMARY:
The purpose of this study is to test the effectiveness of physician profiling and care coordination by a diabetes resource nurse in improving the quality of diabetes care.

DETAILED DESCRIPTION:
HealthTexas Provider Network primary care practices with at least 10 Medicare diabetes patients over the age of 65 were randomized to one of 3 intervention arms: physician feedback of process measures using Medicare claims data ("Claims"); feedback of Medicare claims data plus clinical measures from medical record abstraction ("Claims+MR"); or both types of feedback plus a practice-based DRN ("DRN"). For the 12 months prior to the intervention and 12 months post-intervention, performance data on diabetes related processes of care (annual HbA1c testing, annual LDL cholesterol screening, annual hypertension screening, annual eye, foot, and renal assessment) and patient outcomes (HbA1c level, LDL cholesterol level, blood pressure) were collected from medical record abstraction and Medicare claims data. Pre-post change scores will be compared between intervention arms to examine effectiveness of physician profiling and care coordination by a diabetes resource nurse.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 65 years on January 1, 2000
* diagnosis of diabetes mellitus
* diabetes related visit to HTPN physician within the past year
* Resident of Texas
* Medicare insurance coverage

Exclusion Criteria:

* Patient chart not available for abstraction

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1891 (Actual)
Dates: Start 2000-01; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Ballard, MD,MSPH,PhD, Principal Investigator — Baylor Health Care System Institute for Health Care Research and Improvement
Locations (1):
- Baylor Health Care System Institute for Health Care Research and Improvement, Dallas, Texas, United States

REFERENCES:
- [Result] Hollander P, Nicewander D, Couch C, Winter D, Herrin J, Haydar Z, Ballard DJ. Quality of care of Medicare patients with diabetes in a metropolitan fee-for-service primary care integrated delivery system. Am J Med Qual. 2005 Nov-Dec;20(6):344-52. doi: 10.1177/1062860605280205. PMID 16280398
- [Result] Herrin J, Nicewander DA, Hollander PA, Couch CE, Winter FD, Haydar ZR, Warren SS, Ballard DJ. Effectiveness of diabetes resource nurse case management and physician profiling in a fee-for-service setting: a cluster randomized trial. Proc (Bayl Univ Med Cent). 2006 Apr;19(2):95-102. doi: 10.1080/08998280.2006.11928137. PMID 16609732

RESULTS

PARTICIPANT FLOW:
Groups:
- Claims: Physician feedback of patient process measures using Medicare claims data
- Claims+MR: Physician feedback of patient process measures using Medicare claims data plus medical record-abstracted clinical measures
- Claims+MR+Diabetes Resource Nurse: Physician Feedback of patient process measures using Medicare claims data and medical record-abstracted clinical measures, plus patient access to a diabetes resource nurse.
Period: Overall Study
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Started | 597 | 811 | 602
Completed | 565 | 758 | 568
Not Completed | 32 | 53 | 34
Not completed — Death | 32 | 53 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse | Total
Number analyzed (Participants) | 565 | 758 | 568 | 1891
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 565 | 758 | 568 | 1891
Age, Continuous [Mean (Standard Deviation); unit: years] — Patient characteristics were only described by study arm for the 1891 patients who survived to final follow-up.
  years | 73.1 (0.1) | 72.6 (0.1) | 73.2 (0.1) | 72.9 (0.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Patient characteristics were only calculated by study arm for the 1891 patients who survived to final follow-up.
  Participants
    Female | 290 | 380 | 279 | 949
    Male | 275 | 378 | 289 | 942
number of patients with HbA1c <9 percent [Number; unit: participants] — This measure reports the number of patients in each study arm who had achieved the recommended level of glycemic control, as demonstrated by an HbA1c value of <9%. As not all patients achieved this level of control, the numbers differ from the Overall Number of Baseline Participants.
  participants | 461 | 630 | 481 | 1572
Number of patients with LDL cholesterol <100mg/dL [Number; unit: participants] — This measure reports the number of patients in each study arm who had achieved the recommended level of LDL cholesterol control, as demonstrated by value <100 mg/dL. As not all patients achieved this level of control, the numbers differ from the Overall Number of Baseline Participants.
  participants | 158 | 244 | 198 | 600
Number of patients with blood pressure <130/80 mmHg [Number; unit: participants] — This measure reports the number of patients in each study arm who had achieved the recommended level of blood pressure control, as demonstrated by a value <130/80 mmHg. As not all patients achieved this level of control, the numbers differ from the Overall Number of Baseline Participants.
  participants | 110 | 136 | 99 | 345
Mean HbA1c level [Mean (Standard Deviation); unit: percent] | 7.2 (1.5) | 7.2 (1.4) | 7.1 (1.4) | 7.2 (0.03)
mean LDL level [Mean (Standard Deviation); unit: mg/dL] | 106.9 (32.9) | 104.6 (32.6) | 104.3 (33.9) | 104.9 (0.9)
mean diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 76.0 (9.9) | 77.7 (9.5) | 77.1 (9.8) | 76.8 (0.2)
mean systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 139.5 (18.5) | 139.7 (18.6) | 140.2 (18.0) | 139.6 (0.4)
number of patients with annual HbA1c assessment (as determined from medical record review) [Number; unit: participants] — Not all patients had an HbA1c test documented in the medical record within the past 12 months. As such, the number of participants in each study arm that have an annual HbA1c assessment is lower than the total number of baseline participants in that study arm.
  participants | 508 | 693 | 562 | 1763
Number of patients with an annual lipid assessment (as determined from medical record review) [Number; unit: participants] — As not all patients had a lipid assessment documented in the medical record for the previous 12 months, the number of patients reported in each study arm for this measure is lower than the total number of baseline participants in that study arm.
  participants | 380 | 567 | 441 | 1388
Number of patients with annual blood pressure assessment (as determined from medical record review) [Number; unit: participants] — As not all patients had a blood pressure assessment documented in the medical record for the previous 12 months, the number of patients reported in each study arm for this measure is lower than the total number of baseline participants in that study arm.
  participants | 562 | 751 | 561 | 1874
Number of patients with an annual eye exam (as determined from medical record review) [Number; unit: participants] — As not all patients had an eye assessment documented in the medical record for the previous 12 months, the number of patients reported in each study arm for this measure is lower than the total number of baseline participants in that study arm.
  participants | 61 | 127 | 119 | 307
Number of patients with an annual foot exam (as determined from medical record review) [Number; unit: participants] — As not all patients had an eye exam documented in the medical record for the previous 12 months, the number of patients reported in each study arm for this measure is lower than the total number of baseline participants in that study arm.
  participants | 229 | 409 | 363 | 1001
Number of patients with annual renal function test (as determined from medical record review) [Number; unit: participants] — As not all patients had a renal function test documented in the medical record for the previous 12 months, the number of patients reported in each study arm for this measure is lower than the total number of baseline participants in that study arm.
  participants | 168 | 304 | 234 | 706
Number of patients with annual HbA1c assessment (as determined from Medicare claims data) [Number; unit: participants] — As not all patients had a claim history for an HbA1c test in the previous 12 months, the number of patients reported in each study arm for this measure is lower than the total number of baseline participants in that study arm.
  participants | 512 | 680 | 533 | 1725
Number of patients with an annual eye exam (as determined from Medicare claims data) [Number; unit: participants] — As not all patients had a claim history for an eye exam in the previous 12 months, the number of patients reported in each study arm for this measure is lower than the total number of baseline participants in that study arm.
  participants | 350 | 497 | 353 | 1200
Number of patients with an annual lipid assessment (as determined from Medicare claims data) [Number; unit: participants] — As not all patients had a claim history for a lipid assessment in the previous 12 months, the number of patients reported in each study arm for this measure is lower than the total number of baseline participants in that study arm.
  participants | 398 | 582 | 448 | 1428
Number of patients with a semi-annual HbA1c assessment (as determined form Medicare claims data) [Number; unit: participants] — As not all patients had claims histories for 2 HbA1c tests in the previous 12 months, the number of patients reported in each study arm for this measure is lower than the total number of baseline participants in that study arm.
  participants | 394 | 540 | 434 | 1368

OUTCOME MEASURES:

1. Primary Outcome: Change Score for "HbA1c <9 Percent"
Description: Each patient was assigned a "change score" of -1, 0, or 1. A positive value indicated a patient non-adherent to the guideline recommendation for HbA1c <9 percent at baseline had achieved such a level at follow up. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: This measure compared baseline values (01/01/2000-12/31/2000) to follow-up values (01/01/2001-12/31/2001)
Population: Patients missing either baseline or follow-up values for HbA1c were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 425 | 584 | 437
units on a scale | 0.01 (0.34) | 0.02 (0.32) | 0.04 (0.32)
Statistical Analysis 1: Comparison: Claims vs Claims+MR+Diabetes Resource Nurse; We used a three-stage hierarchical model estimate the effect of the interventions on the change in endpoint from baseline to follow-up. Change scores for dichotomous measures were scored as -1, 0, or 1, with a positive value indicating increased guideline adherence or increased incidence of that process. We used ordered logistic models to test the hypothesis that patients in the intervention groups were more likely to meet guidelines or to receive these processes of care; Test type: Superiority or Other; p = 0.307, Regression, Logistic; Mean Difference (Final Values) = 0.03

2. Primary Outcome: Change Score for "LDL <100 mg/dL"
Description: Each patient was assigned a "change score" of -1, 0, or 1. A positive value indicated that a patient non-adherent to the guideline recommendation of LDL <100 mg/dL at baseline had achieved adherence at follow-up. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (01/01/2000-12/31/2000) to follow-up (01/01/2001-12/31/2001)
Population: Patients missing either baseline or follow-up LDL values were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 268 | 406 | 320
units on a scale | -0.01 (0.52) | 0.07 (0.50) | 0.02 (0.52)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.551, Regression, Logistic; Mean Difference (Final Values) = 0.03

3. Primary Outcome: Change Score for "Blood Pressure (b.p.) <130/80 mmHg"
Description: Each patient was assigned a change score of -1, 0, or 1. A positive value indicated that a patient non-adherent to the guideline recommendation of blood pressure <130/80 mmHg at baseline had achieved adherence at follow-up. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (01/01/2000-12/31/2000) to follow-up (01/01/200112/31/2001)
Population: Patients missing either a baseline or follow-up blood pressure value were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 510 | 680 | 512
units on a scale | 0.05 (0.47) | 0.03 (0.50) | 0.04 (0.45)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.927, Regression, Logistic; Mean Difference (Final Values) = -0.01

4. Secondary Outcome: Change Score for "HbA1c Level"
Description: Change score was calculated by subtracting the follow-up HbA1c value from the baseline value for each patient. Patients missing either a baseline or follow-up value were excluded. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients missing either a baseline or follow-up HbA1c value were excluded.
Measure: Mean (Standard Deviation); unit: change in percentage of glycosolated-Hb
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 425 | 584 | 437
change in percentage of glycosolated-Hb | 0.05 (1.28) | 0.16 (1.44) | 0.14 (1.24)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.308, Regression, Logistic; Mean Difference (Final Values) = 0.09

5. Secondary Outcome: Change Score for "Diastolic Blood Pressure"
Description: Change score was calculated by subtracting the follow-up value from the baseline value for each patient. Patients missing either a baseline or follow-up value were excluded. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients missing either a baseline or follow-up blood pressure measurement were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 510 | 680 | 512
mmHg | 1.21 (10.51) | 1.04 (10.32) | 1.26 (11.73)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.867, Regression, Logistic; Mean Difference (Final Values) = 0.05

6. Secondary Outcome: Change Score for "LDL Level"
Description: Change score was calculated by subtracting the follow-up LDL value from the baseline value for each patient. Patients missing either a baseline or follow-up value were excluded. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients missing either baseline or follow-up LDL values were excluded.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 268 | 406 | 320
mg/dL | 0.22 (28.15) | 3.88 (28.54) | -1.20 (30.37)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.807, Regression, Logistic; Mean Difference (Final Values) = -0.98

7. Secondary Outcome: Change Score for "Systolic Blood Pressure"
Description: as for outcome 5
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients missing either a baseline or follow-up blood pressure measurement were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 510 | 680 | 512
mmHg | 2.35 (20.11) | 1.08 (20.99) | 1.80 (19.97)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.702, Regression, Logistic; Mean Difference (Final Values) = -0.55

8. Secondary Outcome: Change Score for "Annual HbA1c Assessment" (as Determined From Medical Record Review)
Description: Each patient was assigned a change score of -1, 0, or 1. A positive value indicated a patient who was non-compliant with the guideline recommendation for an annual HbA1c assessment in the baseline period was compliant in the follow-up period. Patients missing either a baseline or follow-up value were excluded. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients for whom records were missing for either baseline or follow-up were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 564 | 758 | 566
units on a scale | -0.08 (0.45) | -0.09 (0.44) | -0.10 (0.45)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.413, Regression, Logistic; Mean Difference (Final Values) = -0.02

9. Secondary Outcome: Change Score for "Annual Lipid Assessment" (as Determined From Medical Record Review)
Description: Each patient was assigned a change score of -1, 0, or 1. A positive value indicated a patient who was non-compliant with the guideline recommendation for an annual lipid assessment in the baseline period was compliant in the follow-up period. Patients missing either a baseline or follow-up value were excluded. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients for whom either baseline or follow-up records were missing were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 564 | 758 | 566
units on a scale | 0.00 (0.55) | -0.06 (0.52) | -0.01 (0.53)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.996, Regression, Logistic; Mean Difference (Final Values) = -0.01

10. Secondary Outcome: Change Score for "Annual Blood Pressure Assessment" (as Determined From Medical Record Review)
Description: Each patient was assigned a change score of -1, 0, or 1. A positive value indicated a patient who was non-compliant with the guideline recommendation for an annual blood pressure assessment in the baseline period was compliant in the follow-up period. Patients missing either a baseline or follow-up value were excluded. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients for whom either baseline or follow-up records were missing were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 564 | 758 | 566
units on a scale | -0.09 (0.29) | -0.09 (0.30) | -0.07 (0.30)
Statistical Analysis 1: Comparison: Claims vs Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.451, Regression, Logistic; Median Difference (Final Values) = 0.02

11. Secondary Outcome: Change Score for "Annual Foot Exam" (as Determined by Medical Record Review)
Description: Each patient was assigned a change score of -1, 0, or 1. A positive value indicated a patient who was non-compliant with the guideline recommendation for an annual foot exam in the baseline period was compliant in the follow-up period. Patients missing either a baseline or follow-up value were excluded. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients for whom baseline or follow-up records were not available were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 564 | 758 | 566
units on a scale | -0.11 (0.56) | -0.06 (0.67) | -0.01 (0.59)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.447, Regression, Logistic; Median Difference (Final Values) = 0.10

12. Secondary Outcome: Change Score for "Annual Eye Exam" (as Determined From Medical Record Review)
Description: Each patient was assigned a change score of -1, 0, or 1. A positive value indicated a patient who was non-compliant with the guideline recommendation for an annual eye exam in the baseline period was compliant in the follow-up period. Patients missing either a baseline or follow-up value were excluded. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients for whom records were not available at either baseline or follow-up were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 564 | 758 | 566
units on a scale | -0.01 (0.37) | -0.02 (0.46) | 0.00 (0.52)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.936, Regression, Logistic; Median Difference (Final Values) = 0.01

13. Secondary Outcome: Change Score for "Annual Renal Function Assessment" (as Determined From Medical Record Review)
Description: Each patient was assigned a change score of -1, 0, or 1. A positive value indicated a patient who was non-compliant with the guideline recommendation for an annual renal function assessment in the baseline period was compliant in the follow-up period. Patients missing either a baseline or follow-up value were excluded. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients for whom records were not available at either baseline or follow-up were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 564 | 758 | 566
units on a scale | 0.04 (0.48) | 0.07 (0.49) | 0.08 (0.46)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.332, Regression, Logistic — A comparison of the claims vs. claims+MR arms was also conducted, giving a p-value of 0.537; Median Difference (Final Values) = 0.04

14. Secondary Outcome: Change Score for "Annual HbA1c Assessment" (as Determined From Medicare Claims Data)
Description: as for outcome 8
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients for whom records were not available at either baseline or follow-up were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 564 | 758 | 566
units on a scale | -0.16 (0.51) | -0.16 (0.51) | -0.17 (0.47)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.860, Regression, Logistic; Median Difference (Final Values) = -0.01

15. Secondary Outcome: Change Score for "Annual Eye Exam" (as Determined From Medicare Claims Data)
Description: as for outcome 12
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients for whom records were not available at either baseline or follow-up were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 564 | 758 | 566
units on a scale | -0.09 (0.54) | -0.06 (0.59) | -0.06 (0.54)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.382, Regression, Logistic; Mean Difference (Final Values) = 0.03

16. Secondary Outcome: Change Score for "Annual Lipid Assessment" (as Determined From Medicare Claims Data)
Description: as for outcome 9
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients for whom records were not available at either baseline or follow-up were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 564 | 758 | 566
units on a scale | -0.09 (055) | -0.15 (0.57) | -0.08 (0.53)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.988, Regression, Logistic; Mean Difference (Final Values) = 0.01

17. Secondary Outcome: Change Score for "Semiannual HbA1c Assessment" (as Determined From Medicare Claims Data)
Description: Each patient was assigned a change score of -1, 0, or 1. A positive value indicated a patient who was non-compliant with the guideline recommendation for a semi-annual HbA1c assessment in the baseline period was compliant in the follow-up period. Patients missing either a baseline or follow-up value were excluded. Patient-level change scores were then summed and averaged over each study arm.
Time Frame: change from baseline (1/1/2000-12/31/2000) to follow-up (1/1/2001-12/31/2001)
Population: Patients for whom records were not available at either baseline or follow-up were excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Number analyzed (Participants) | 564 | 758 | 566
units on a scale | -0.12 (0.62) | -0.11 (0.62) | -0.11 (0.56)
Statistical Analysis 1: Comparison: Claims+MR+Diabetes Resource Nurse; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.685, Regression, Logistic; Mean Difference (Final Values) = 0.01

ADVERSE EVENTS:
Time Frame: This study was conducted from 1/1/2000-12/31/2001. All the interventions tested were at the practice level and did not directly impact patient care. Since patients were receiving 'usual care', no adverse event data were collected.
Description: The interventions tested were all tools/resources to help practices improve performance on diabetes quality measures. All decisions about patient treatment remained with the individual physicians, at their discretion. Thus, patients were not placed at additional risk through the practices' participation in the study, and adverse events not tracked.
Arm/Group | Claims | Claims+MR | Claims+MR+Diabetes Resource Nurse
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
All participating practices belonged to the same network of fee-for-service practices, which may reduce generalizability.

Neither physicians nor patients could be blinded; but data were collected by individuals blinded to study arm assignments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No